CLINICAL TRIAL: NCT02590575
Title: "Low Flow" CO2 Removal Via a Membrane Gas Exchange Device (Prismalung®) on a Renal Replacement Platform (Prismaflex®) in Hypercapnic, Ventilated Patients Requiring Renal Replacement
Brief Title: "Low Flow" CO2 Removal on RRT
Acronym: Prismalung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Goethe University (Other)
Responsible Party: Principal Investigator, stefan john, Prof. Dr. med. Stefan John, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ_G_023.14-II-4
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Renal Replacement Therapy
Keywords: extracorporeal CO2 removal; renal replacement therapy; Prismalung; ARDS; hypercapnia; Changes in the arterial pCO2 value; ventilated; Hypercapnic
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CO2 removal (Other)
  Interventions: Device: Extracorporeal CO2 removal with the Prismalung(R) gas exchanger on the Prismaflex(R) renal replacement platform

INTERVENTIONS:
Device: Extracorporeal CO2 removal with the Prismalung(R) gas exchanger on the Prismaflex(R) renal replacement platform — 1. With ongoing continuous hemofiltration and mechanical ventilation additional membrane gas exchange device (Prismalung®) in the renal replacement circulation; measurements of the effects on PaCO2 under varying blood and sweep gas flows
  2. Afterwards, reduction of the tidal volume (VT) / plateau pressure until reaching the initial PaCO2value

SUMMARY:
The purpose of this study is to test the effectiveness of a membrane gas exchange device in the venovenous circulation of a continuous renal replacement therapy for the purpose of CO2 elimination and pH compensation. Thus, the primary endpoint is the modification of the PaCO2 and/or the ventilator settings (tidal volume VT and plateau pressure Pplat).

DETAILED DESCRIPTION:
Protocol synopsis Study title "Low flow" CO2 removal via a membrane gas exchange device (Prismalung®) on a renal replacement platform (Prismaflex®) in hypercapnic, ventilated patients requiring renal replacement therapy Brief description Prismalung Study Indication Hypercapnic, ventilated, and renal replacement therapy requiring patients Primary study goal Changes in the arterial pCO2 value Secondary study goals Changes in the acid-base balance Changes of tidal volumes/ventilation pressures Changes in hemodynamics Study design Prospective intervention study (pilot study)

Study population Inclusion criteria:

1. Necessity of renal replacement therapy
2. Necessity of ventilation therapy with an expected duration >24 hrs. in mild to moderate ARDS according to the "Berlin Definition" (300≥PaO2/FiO2>100mmHg, ventilated acc. to the ARDS network strategy with VT 6 ml/kgKG (KG = Körpergewicht, body weight) and PEEP ≥ 5 cmH2O)Pneumonia, pulmonary vasculitis, COPD, or other pulmonary disorder
3. PaCO2 ≥ 55 mmHg with plateau ventilation pressure > 25 cmH2O and pH < 7.30
4. Written consent by patient or legal representative

Number of patients n = 20 Interventions 1. With ongoing continuous hemofiltration and mechanical ventilation additional membrane gas exchange device (Prismalung®) in the renal replacement circulation; measurements of the effects on PaCO2 under varying blood and sweep gas flows 2. Afterwards, reduction of the tidal volume (VT) / plateau pressure until reaching the initial PaCO2value Study drug None Primary endpoint 1. Changes in the PaCO2 / acid-base status (BGA) 2. Changes of the VT / plateau pressure in the ventilation (ventilation settings) Secondary endpoints Changes in the systemic hemodynamics Vasopressor dosage BGA, renal values, lactate PaCO2 before and after gas exchange device Lifetimes of the extracorporeal circulation Complications Study site Intensive care units Medizinische Klinik 4, Uniklinikum Erlangen-Nürnberg Medizinische Klinik 4, Klinikum Nürnberg Süd Klinik für Intensivmedizin Universitätsklinikum Hamburg Eppendorf Klinik für Anästhesiologie und Intensivmedizin Universitätsklinikum Frankfurt a. M. Timeline Start in October 2015 Anticipated study duration: 6 months Financing Baxter Gambro Renal GmbH (Ltd)

ELIGIBILITY:
Inclusion Criteria:

1. Necessity of renal replacement therapy
2. Necessity of ventilation therapy with an expected duration >24 hrs. in mild to moderate ARDS according to the "Berlin Definition" (300≥PaO2/FiO2>100mmHg, ventilated acc. to the ARDS network strategy with VT 6 ml/kgKG (KG = Körpergewicht, body weight) and PEEP ≥ 5 cmH2O) Pneumonia, pulmonary vasculitis, COPD, or other pulmonary disorder
3. PaCO2 ≥ 55 mmHg with plateau ventilation pressure > 25 cmH2O and pH < 7.30
4. Written consent by patient or legal representative

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. BMI > 40 kg/m2
4. Decompensated heart failure or acute stroke
5. Severe ARDS (PaO2/FiO2 < 100 mmHg)
6. Acute cranio-cerebral injury
7. Severe liver failure (Child-Pugh score >7)
8. Heparin-induced thrombopenia (HIT II)
9. Contraindications to the performance of CVVH (continuous venovenous hemofiltration)
10. Contraindications to systemic anticoagulation
11. Lacking possibility of access via a dialysis catheter
12. Surgeries scheduled within 48 hrs of inclusion in the study
13. Advanced tumor disorder with life expectancy < 1 month
14. Moribund patients, decision to forego therapy
15. Lacking consent
16. Participation in a different intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in the PaCO2, acid-base status (BGA) | hours to 3 days
Changes of the VT / plateau pressure in the ventilation (ventilation settings) | hours to 3 days

SECONDARY OUTCOMES:
Changes in mean arterial pressure (mmHg) | hours to 3 days
Changes in heart rate (bpm) | hours to 3 days
Changes in norepinephrin dose (mg/h) | hours to 3 days
Changes in Serum lactate concentration (mmol/l) | hours to 3 days
Arterial pO2 and pCO2 (mmHg) | hours to 3 days
Arterial bicarbonate concentration (mmol/l) | hours to 3 days
Standard Base Excess (mmol/l) | hours to 3 days
Changes in Serum creatinine (mg/dl) | hours to 3 days
PCO2 before and after gas exchange device (mmHg) | hours to 3 days
Lifetime of extracorporeal circuit in hours (Duration from start to end of RRT) | hours to 3 days
Number and kind of adverse events during study period deemed clinically significant by investigator (as documented by paper questionnaire) | hours to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan John, MD, Principal Investigator — University of Erlangen-Nuernberg
Locations (1):
- University of Erlangen-Nuernberg, Nuremberg, Germany

REFERENCES:
- [Derived] Nentwich J, Wichmann D, Kluge S, Lindau S, Mutlak H, John S. Low-flow CO2 removal in combination with renal replacement therapy effectively reduces ventilation requirements in hypercapnic patients: a pilot study. Ann Intensive Care. 2019 Jan 7;9(1):3. doi: 10.1186/s13613-019-0480-4. PMID 30617611